CLINICAL TRIAL: NCT03824314
Title: Comparison of the Effect of Adding Midazolam Versus Fentanyl to Intrathecal Levobupivacaine in Patients Undergoing Caesarean Section
Brief Title: Effect of Adding Midazolam Versus Fentanyl to Intrathecal Levobupivacaine in Patients Undergoing Caesarean Section
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mohamed Abdelrady Mohamed (Other)
Responsible Party: Sponsor-Investigator, Mohamed Abdelrady Mohamed, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: midazolam versus fentanyl
Record Dates: First submitted 2019-01-19; First posted 2019-01-31 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-05

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Experimental): . Group M (n = 40) receive 2 ml of 0.5% isobaric levobupivacaine (10 mg) plus 0.5 ml midazolam (2 mg) ) intrathecally
  Interventions: Drug: Midazolam
- group F (Experimental): group F (n = 40) receive 2 ml of 0.5% isobaric levobupivacaine (10 mg) plus 0.5 ml fentanyl (25 μg) intrathecally.
  Under all aseptic precautions, spinal anaesthesia will be given in L3 and L4 space with 25 gauge Quincke spinal needle via midline approach in sitting position. On free flow of cerebrospinal fluid, study drug will be injected intrathecally . Patients will immediately turn to supine position
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Midazolam — 2 ml of 0.5% isobaric levobupivacaine (10 mg) plus 0.5 ml midazolam (2 mg)will be given intrathecally in L3 and L4 space with 25 gauge Quincke spinal needle via midline approach in sitting position. On free flow of cerebrospinal fluid, study drug will be injected intrathecally . Patients will immediately turn to supine position
  Arms: Group M
Drug: Fentanyl — 2 ml of 0.5% isobaric levobupivacaine (10 mg) plus 0.5 ml fentanyl (25 μg)will be given intrathecally in L3 and L4 space with 25 gauge Quincke spinal needle via midline approach in sitting position. On free flow of cerebrospinal fluid, study drug will be injected intrathecally . Patients will immediately turn to supine position
  Arms: group F

SUMMARY:
The aim of this study is to compare the effects of intrathecal levobupivacaine plus midazolam and levobupivacaine plus fentanyl in patients undergoing caesarean section to get a prolonged postoperative analgesic effect and less side effects

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anaesthesiologists grades I and II ,

Exclusion Criteria:

* pre-existing neurological or spinal disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
1st post-operative analgesic request | 24-hour
  pain will be evaluated using VAS score, every 30 min for 180 min then hourly for 12 h and thereafter every 3 hourly till 24 h of surgery in both groups. Rescue analgesia in the form of injection Ketorolac 30mg I.V when VAS >3 in both groups.

SECONDARY OUTCOMES:
duration of sensory block Total analgesic consumption | 24-hour
  total duration of sensory block (regression to S1 dermatome) will be noted

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No